CLINICAL TRIAL: NCT00420849
Title: A Multicentre, Single-arm, Open-label Safety Study of Lenalidomide Plus Dexamethasone in Previously Treated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-018; 2006-002517-12 (EudraCT Number)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2012-03-14 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

ARMS (1):
- Lenalidomide plus Dexamethasone (Experimental): Lenalidomide administered orally, 25 mg daily (QD) for the first 21 days of each 28-day cycle. Pulse dexamethasone administered orally, 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle during Cycles 1 to 4 (approximately months 1-4). Beginning with Cycle 5 (approximately month 5), a maintenance dose of dexamethasone (40 mg QD) was administered on Days 1 to 4 of each 28-day cycle.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Oral lenalidomide at a dose of 25 mg daily for 21 days every 28 days. Treatment as tolerated until disease progression, drug became commercially available or limited to 6 treatment cycles.
  Other Names: Revlimid
Drug: Dexamethasone — Oral pulse dexamethasone at a dose of 40 mg daily on days 1-4, 9-12, and 17-20 for each 28-day-cycle for cycles 1 through 4. Beginning cycle 5, a maintenance dose of dexamethasone (40 mg QD) was administered on Days 1 to 4 of each 28-day cycle.

SUMMARY:
This is a multi-centre, single-arm treatment study combining lenalidomide plus high dose dexamethasone.

Subjects who qualify for participation will receive lenalidomide plus high dose dexamethasone in 4 week cycles. Subjects will be seen every 2 weeks for the first 3 cycles of therapy and then every 4 weeks after the third cycle until disease progression is documented, study drug is discontinued for any reason or lenalidomide becomes commercially available for this indication. Assessments of safety and quality of life are performed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with multiple myeloma that is progressing after at least 2 cycles of anti-myeloma treatment or that has relapsed with progressive disease after treatment.
* Subjects must discontinue all anti-myeloma drug or non-drug therapy prior to the first dose of study drug with the exception of radiation therapy initiated prior to baseline.
* Females of childbearing potential must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence.

Exclusion Criteria:

* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Therapeutic Area Head
Locations (5):
- The Mater Private Centre for Haematology & Oncology, South Brisbane, Australia
- Wilhelminenspital, Vienna, Montlearstrasse 37, Austria
- St James's Hospital, Dublin, Ireland
- H. Clínico de Salamanca, Salamanca, Spain
- Royal Free Hospital & Medical School, London, United Kingdom

REFERENCES:
- [Result] Yong K, Alegre Amor A, Browne P, Cavenagh J, Dodds T, Greil R, et al. A Multicenter, Single-arm, Open-label Safety and Quality of Life Study of Lenalidomide plus Dexamethasone in previously treated Patients with Multiple Myeloma. Haematologica 2010;95(suppl.2):392, abs. 0944.
- [Derived] Alegre A, Oriol-Rocafiguera A, Garcia-Larana J, Mateos MV, Sureda A, Martinez-Chamorro C, Cibeira MT, Aguado B, Knight R, Rosettani B. Efficacy, safety and quality-of-life associated with lenalidomide plus dexamethasone for the treatment of relapsed or refractory multiple myeloma: the Spanish experience. Leuk Lymphoma. 2012 Sep;53(9):1714-21. doi: 10.3109/10428194.2012.662643. Epub 2012 Mar 1. PMID 22292853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide Plus Dexamethasone
Started | 587
Completed | 256 (Participants completed the study upon commercial availability of lenalidomide)
Not Completed | 331
Not completed — Lack of Efficacy | 154
Not completed — Adverse Event | 107
Not completed — Withdrawal by Subject | 28
Not completed — Death | 18
Not completed — Other | 14
Not completed — Transplant | 8
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.74)
Age, Customized [Number; unit: participants]
  <=18 years | 0
  >18 and <=65 years | 314
  >65 years | 273
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241
  Male | 346
Race/Ethnicity, Customized [Number; unit: participant]
  White | 548
  Other | 17
  Asian / Pacific Islander | 10
  Black | 9
  Hispanic | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence of Treatment-emergent Adverse Events (TEAEs), by Severity, Seriousness, and Relationship to Treatment
Description: Counts of study participants who had treatment-emergent adverse events (TEAEs) defined as any reported AE that started on or after the first day of study drug dosing. A participant with multiple occurrences of an adverse event within a category is counted only once in that category.
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) was used by investigators to assess TEAEs. Severity scale ranges from 0 (none) to 5 (death). Grade 3=severe AE; Grade 4=life threatening or disabling AE; Grade 5=death.
Time Frame: up to 123 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
participants
  At least one treatment-emergent AE (TEAE) | 586
  At least one TEAE related to study drug | 519
  At least one TEAE with severity grade of 3 or 4 | 471
  At least one serious AE (SAE) | 340

2. Secondary Outcome: Participants With Adverse Events of Special Interest: Peripheral Neuropathy
Description: Number of participants with at least one peripheral neuropathy treatment-emergent adverse event (TEAE), and number of participants reporting AEs coded to preferred terms that comprise the search terms for peripheral neuropathy in MedDRA version 9.0 are listed. A participant with multiple occurrences of a TEAE was counted only once for that category.
Time Frame: up to 124 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
participants
  At least one TEAE of peripheral neuropathy | 84
  Neuropathy peripheral | 46
  Peripheral sensory neuropathy | 33
  Neuralgia | 5
  Peripheral motor neuropathy | 2
  Polyneuropathy | 2
  Sensory disturbance | 1

3. Secondary Outcome: Time to First Peripheral Neuropathy Treatment-Emergent Adverse Event (TEAE)
Description: Time between first dose and when a TEAE for peripheral neuropathy was reported. The mean is the univariate mean without adjusting for censoring. The treatment duration was used for censored participants.
Time Frame: up to 124 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
weeks | 25.6 (21.53)

4. Secondary Outcome: Participants With Adverse Events of Special Interest: Venous Thromboembolic Events
Description: Number of participants with at least one venous thromboembolic treatment-emergent adverse event (TEAE), and number of participants reporting AEs coded to preferred terms that comprise the search terms for venous thromboembolic events in MedDRA version 9.0 are listed. A participant with multiple occurrences of a TEAE was counted only once for that category.
Time Frame: up to 124 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
participants
  At least one venous thromboembolic event | 60
  Deep vein thrombosis | 38
  Pulmonary embolism | 23
  Thrombophlebitis | 7
  Venous thrombosis limb | 1

5. Secondary Outcome: Time to First Venous Thromboembolic Treatment-Emergent Adverse Event (TEAE)
Description: Time between first dose and when a TEAE for venous thromboembolic event was reported. The mean is the univariate mean without adjusting for censoring. The treatment duration was used for censored participants.
Time Frame: up to 124 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 587
weeks | 26.5 (21.51)

6. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Physical Functioning Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lenalidomide - Subpopulation From Austria + Australia: Lenalidomide administered orally, 25 mg daily (QD) for the first 21 days of each 28-day cycle. Pulse dexamethasone administered orally, 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle during Cycles 1 to 4 (approximately months 1-4). Beginning with Cycle 5 (approximately month 5), a maintenance dose of dexamethasone (40 mg QD) was administered on Days 1 to 4 of each 28-day cycle. Subpopulation includes participants from Austria and Australia
- Lenalidomide - Subpopulation From UK + Ireland: Lenalidomide administered orally, 25 mg daily (QD) for the first 21 days of each 28-day cycle. Pulse dexamethasone administered orally, 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle during Cycles 1 to 4 (approximately months 1-4). Beginning with Cycle 5 (approximately month 5), a maintenance dose of dexamethasone (40 mg QD) was administered on Days 1 to 4 of each 28-day cycle. Subpopulation includes participants from the UK and Ireland.
- Lenalidomide - Subpopulation From Spain: Lenalidomide administered orally, 25 mg daily (QD) for the first 21 days of each 28-day cycle. Pulse dexamethasone administered orally, 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle during Cycles 1 to 4 (approximately months 1-4). Beginning with Cycle 5 (approximately month 5), a maintenance dose of dexamethasone (40 mg QD) was either administered on Days 1 to 4 of each 28-day cycle or on Days 1, 8, 15, and 22 of each 28-day cycle. Subpopulation includes participants from Spain.
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 153 | 123 | 38
units on a scale | -3.6 (16.19) | -2.9 (16.54) | -1.8 (15.10)

7. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Role Functioning Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of role functioning.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 122 | 38
units on a scale | -2.4 (26.05) | -1.5 (32.50) | -2.6 (31.61)

8. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Emotional Functioning Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of emotional functioning.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 151 | 123 | 38
units on a scale | -0.2 (15.92) | -4.0 (19.17) | -0.7 (27.32)

9. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Cognitive Functioning Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of cognitive functioning.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 123 | 38
units on a scale | -1.9 (19.61) | -4.9 (23.06) | 3.5 (16.96)

10. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Social Functioning Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better level of social functioning.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 123 | 38
units on a scale | -5.2 (26.25) | -5.3 (29.67) | -3.1 (30.72)

11. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the fatigue scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 123 | 38
units on a scale | 2.6 (20.93) | 5.3 (26.59) | 1.0 (22.07)

12. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Pain Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the pain scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 153 | 125 | 38
units on a scale | -3.9 (25.56) | -5.2 (28.35) | -6.6 (32.77)

13. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Nausea/Vomiting Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the nausea/vomiting scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 123 | 38
units on a scale | 1.0 (13.99) | 0.1 (17.14) | -2.2 (19.82)

14. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Constipation Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the constipation scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 150 | 123 | 38
units on a scale | 1.1 (31.71) | 7.9 (26.68) | 2.6 (37.47)

15. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Diarrhea Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the diarrhea scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 151 | 123 | 37
units on a scale | 8.6 (24.18) | 8.1 (24.27) | 9.0 (24.40)

16. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Insomnia Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the insomnia scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 151 | 123 | 37
units on a scale | -3.8 (29.70) | 2.2 (35.38) | -1.8 (34.20)

17. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Dyspnoea Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the dyspnoea scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 148 | 122 | 38
units on a scale | 2.7 (25.94) | 2.7 (27.97) | -0.9 (28.46)

18. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Appetite Loss Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a symptom scale like the appetite loss scale = higher level of symptomatology/problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 123 | 37
units on a scale | 0.4 (27.12) | 3.3 (30.60) | -4.5 (29.57)

19. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Financial Problems Scale
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score for a problem scale like the financial problems scale = higher level of financial problems.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 121 | 38
units on a scale | 2.0 (20.74) | 0.8 (22.14) | 0.9 (16.42)

20. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Quality of Life Scale
Description: EORTQ QLC-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better quality of life.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 152 | 122 | 38
units on a scale | 1.1 (20.90) | -1.8 (23.17) | -2.2 (21.81)

21. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Disease Symptoms Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score for the disease symptoms scale = higher level of symptomatology.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 151 | 122 | 37
units on a scale | -2.4 (16.79) | -1.2 (17.62) | -3.9 (19.00)

22. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Side Effects Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale; higher score for the side effects scale = higher level of symptomatology.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 151 | 121 | 37
units on a scale | 4.9 (13.22) | 4.7 (13.16) | 2.0 (13.45)

23. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Future Perspective Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale. For the future perspective scale, higher score = better perspective of the future.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 150 | 119 | 38
units on a scale | 5.8 (21.14) | 3.4 (21.70) | 4.4 (21.85)

24. Secondary Outcome: Change From Baseline to Week 24 in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Body Image Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. Questions used 4-point scale (1 'Not at All' to 4 'Very Much'). Scores are averaged, and transformed to 0-100 scale. For the body image scale, higher scores = better body image.
Time Frame: Baseline (Day 0), Week 24
Population: Full analysis set of participants who completed the questionnaire at baseline and week 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide - Subpopulation From Austria + Australia | Lenalidomide - Subpopulation From UK + Ireland | Lenalidomide - Subpopulation From Spain
Number analyzed (Participants) | 149 | 117 | 38
units on a scale | -4.3 (35.15) | -2.0 (33.42) | -5.3 (31.51)

ADVERSE EVENTS:
Time Frame: Up to 123 weeks
Description: A participant with multiple occurrences of a serious treatment-emergent adverse event (TEAE) was counted only once for that preferred term.
Arm/Group | Lenalidomide Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 340/587
Other Adverse Events (participants affected / at risk) | 579/587
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=587)
Pneumonia (Infections and infestations) | 52
Lower respiratory tract infection (Infections and infestations) | 38
Sepsis (Infections and infestations) | 17
Respiratory tract infection (Infections and infestations) | 15
Cellulitis (Infections and infestations) | 14
Infection (Infections and infestations) | 7
Neutropenic sepsis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 6
Lobar pneumonia (Infections and infestations) | 5
Septic shock (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 4
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3
Lung infection pseudomonal (Infections and infestations) | 3
Arthritis bacterial (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 2
Febrile infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Abscess oral (Infections and infestations) | 1
Anal infection (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Brain abscess (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis acute (Infections and infestations) | 1
Bronchitis moraxella (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Cellulitis staphylococcal (Infections and infestations) | 1
Central line infection (Infections and infestations) | 1
Cholecystitis infection (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Joint abscess (Infections and infestations) | 1
Legionella infection (Infections and infestations) | 1
Listeria sepsis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Meningitis streptococcal (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Pneumonia moraxella (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Subacute endocarditis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 31
Febrile neutropenia (Blood and lymphatic system disorders) | 22
Neutropenia (Blood and lymphatic system disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Pancytopenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 30
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 6
General physical health deterioration (General disorders) | 4
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 3
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
Drug interaction (General disorders) | 1
Hyperplasia (General disorders) | 1
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Sudden death (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myeloma recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 25
Hypotension (Vascular disorders) | 5
Orthostatic hypotension (Vascular disorders) | 4
Arterial thrombosis limb (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Phlebitis superficial (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Atrial fibrillation (Cardiac disorders) | 12
Cardiac failure (Cardiac disorders) | 7
Acute myocardial infarction (Cardiac disorders) | 4
Angina unstable (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Renal failure acute (Renal and urinary disorders) | 16
Renal failure (Renal and urinary disorders) | 8
Renal impairment (Renal and urinary disorders) | 7
Bladder disorder (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Renal tubular acidosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dizziness (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 3
Syncope vasovagal (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Cranial nerve paralysis (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Phantom pain (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Serotonin syndrome (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Intestinal obstruction (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Tetany (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Fall (Injury, poisoning and procedural complications) | 5
Accidental overdose (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Confusional state (Psychiatric disorders) | 13
Agitation (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 1
Korsakoff's psychosis alcoholic (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Blood creatinine increased (Investigations) | 5
International normalised ratio increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood calcium decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood culture positive (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Steroid withdrawal syndrome (Endocrine disorders) | 2
Hyperparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Oedema genital (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Vision blurred (Eye disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=587)
Fatigue (General disorders) | 249
Neutropenia (Blood and lymphatic system disorders) | 243
Muscle spasms (Musculoskeletal and connective tissue disorders) | 202
Constipation (Gastrointestinal disorders) | 194
Diarrhoea (Gastrointestinal disorders) | 180
Insomnia (Psychiatric disorders) | 173
Anaemia (Blood and lymphatic system disorders) | 154
Thrombocytopenia (Blood and lymphatic system disorders) | 125
Tremor (Nervous system disorders) | 113
Oedema peripheral (General disorders) | 101
Nausea (Gastrointestinal disorders) | 98
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 96
Upper respiratory tract infection (Infections and infestations) | 92
Dizziness (Nervous system disorders) | 87
Muscular weakness (Musculoskeletal and connective tissue disorders) | 84
Back pain (Musculoskeletal and connective tissue disorders) | 83
Rash (Skin and subcutaneous tissue disorders) | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 75
Lethargy (Nervous system disorders) | 74
Headache (Nervous system disorders) | 67
Lower respiratory tract infection (Infections and infestations) | 67
Nasopharyngitis (Infections and infestations) | 64
Dysgeusia (Nervous system disorders) | 63
Pyrexia (General disorders) | 58
Arthralgia (Musculoskeletal and connective tissue disorders) | 56
Vision blurred (Eye disorders) | 55
Mood altered (Psychiatric disorders) | 53
Asthenia (General disorders) | 52
Anorexia (Metabolism and nutrition disorders) | 48
Hyperglycaemia (Metabolism and nutrition disorders) | 48
Vomiting (Gastrointestinal disorders) | 47
Neuropathy peripheral (Nervous system disorders) | 46
Paraesthesia (Nervous system disorders) | 46
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 43
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43
Dyspepsia (Gastrointestinal disorders) | 41
Confusional state (Psychiatric disorders) | 40
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 40
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 39
Hypocalcaemia (Metabolism and nutrition disorders) | 35
Neuropathy (Nervous system disorders) | 35
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 33
Peripheral sensory neuropathy (Nervous system disorders) | 33
Weight decreased (Investigations) | 33
Respiratory tract infection (Infections and infestations) | 32
Dry mouth (Gastrointestinal disorders) | 34
Urinary tract infection (Infections and infestations) | 32
Mouth ulceration (Gastrointestinal disorders) | 31
Shoulder pain (Musculoskeletal and connective tissue disorders) | 31
Bone pain (Musculoskeletal and connective tissue disorders) | 30

LIMITATIONS AND CAVEATS:
This study was defined primarily as an expanded access program in the selected countries. Treatment was to continue until disease progression, study drug was discontinued for any reason, or lenalidomide became commercially available for indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Multicenter publication must include input from investigators and Celgene, agreement to be established before publication. It has priority over subset (single center) publication, for duration of 1 year after study completion.
* Individual investigators have publication right after multicenter publication is complete (or 1 year after study completion), whichever is first. In this case, Celgene has the right to comment and right to ask delay of publication for 180 days.